CLINICAL TRIAL: NCT01994811
Title: Eastern Caribbean Health Outcomes Research Network (ECHORN)
Acronym: ECHORN
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1108008959; 5U24MD006938 (NIH)
Record Dates: First submitted 2013-11-19; First posted 2013-11-26 (Estimated); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Cancer; Cardiovascular Disease; Diabetes
Keywords: cancer; cardiovascular disease; diabetes
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Saliva samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Eastern Caribbean Health Outcomes Research Network (ECHORN) is a collaborative research study that examines the lifestyles, eating habits, and health behaviors associated with cancer, diabetes and heart disease in adult men and women living in the Eastern Caribbean.

DETAILED DESCRIPTION:
The Eastern Caribbean Health Outcomes Research Network (ECHORN) has two aims: (1) To form a research collaborative across the Eastern Caribbean islands of Puerto Rico, the U.S. Virgin Islands, Barbados, and Trinidad & Tobago to recruit and follow a community-dwelling adult cohort to estimate the prevalence of known and potential risk factors associated with the development of heart disease, cancer, and diabetes and (2) To enhance health outcomes research leadership capacity in the region through a series of dedicated activities locally and abroad. ECHORN will expand clinical research with racial/ethnic minority populations in a transitioning part of the globe now threatened with an epidemic of noncommunicable chronic diseases (NCD). ECHORN's findings will have direct implications for the health disparities research and policy agenda in the mainland United States. In the long term, the links ECHORN will facilitate with local health policy delegations and global strategic organizational partners will promote the translation of research to improve health outcomes across the region. The collection and storage of biological specimens will also contribute to national biomonitoring projects and has the potential to identify unique risk and protective factors in the development of NCD.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 40 years of age
* English or Spanish language speaking
* Resident of island at least 10 years
* Able to provide informed consent
* Non-institutionalized at the time of data collection
* Stable contact/residential information
* No plans to relocate from island within the next 5 years

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population-based prospective cohort is comprised of adults aged 40 and older living in four countries: Puerto Rico (PR), Barbados (BB), the US Virgin Islands (USVI), and Trinidad and Tobago (TT).
Sampling Method: Non-Probability Sample
Enrollment: 2961 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
Prevalence of non-communicable diseases | 5 years
  Prevalence of non-communicable diseases, including cancer, heart disease and diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Marcella Nunez-Smith, MD, MHS, Principal Investigator — Yale University
Locations (4):
- University of the West Indies, Cave Hill Campus, Bridgetown, Barbados
- University of Puerto Rico Medical Sciences Campus, San Juan, Puerto Rico
- University of the West Indies, St. Augustine Campus, Saint Augustine, West Indies, Trinidad and Tobago
- University of the Virgin Islands, Charlotte Amalie, Virgin Islands, Virgin Islands

IPD SHARING:
Plan to Share IPD: Yes
A Data Access and Scientific Review Committee (DASR), was been established to oversee requests for research collaboration (e.g. ancillary studies, secondary data analyses, etc.) to ensure they are within the scope of ECHORN's research mandate. Per the ECHORN Data Access Policy, de-identified, limited ECHORN datasets have been made available for public access.
URL: https://www.echorn.org/